CLINICAL TRIAL: NCT05930301
Title: Clinical Research on the Safety and Effectiveness of RT201(Tumor Antigen-specific Macrophage Tumor Vaccine) in the Treatment of Advanced Cervical Cancer
Brief Title: RT201(Tumor Antigen-specific Macrophage Tumor Vaccine)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peihua Lu (Other)
Collaborators: Suzhou Royaltechmed Co.,Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Peihua Lu, Principle Investigator, Wuxi People's Hospital
Organization: Wuxi People's Hospital (Other)
Other Study IDs: WuxiPH
Record Dates: First submitted 2023-06-14; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Cervical
Keywords: Cervical cancer; advanced malignant tumor; Listeria monocytogenes
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single: Mode of administration：IV Administration dosage：10^7/100ml Dosing frequency：Every three weeks

SUMMARY:
This clinical study will include tumor patients in strict accordance with the inclusion and exclusion criteria set in this clinical study, and carry out tumor-specific antigen screening, HLA typing, blood sample collection, cell separation, cell culture and cell reinfusion according to the SOP of Suzhou Ruotai RT201 Cell Therapy. According to the efficacy evaluation criteria set in this clinical study, the included patients will be evaluated and followed up for a long time, and the original data will be saved to provide real and effective clinical data for the safety and efficacy of RT201 tumor single-target individualized clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female patients (≥18 years old);
2. The patient himself voluntarily signed the "informed consent form";
3. HPV positive advanced cervical cancer (refer to FIGO standard);
4. Patients with persistent metastasis or recurrence of squamous cell or non-squamous cell need to be confirmed by histology or cytology;
5. Patients who have received surgical treatment or other standard first-line treatment or patients who cannot receive surgical treatment/chemotherapy/radiotherapy;
6. ECOG≤2
7. Physical condition is good: KPS≥70;
8. The estimated survival time is ≥3 months;
9. Have not received any treatment that may affect the evaluation of curative effect in the past 3 months;
10. The functions of liver, kidney and bone marrow are basically normal: HCT > 25%, white blood cell range 3.5-9.5×109/L, hemoglobin (Hb)≥90g, lymphocyte+monocyte > 20%; Blood Cr≤1.5×UNL (the upper limit of normal) and blood BIL ≤ 1.5× UNL; ALT and AST≤1.5×UNL (for patients with liver metastasis, ALT and ast ≤ 5.0× UNL);
11. Women of childbearing age (15-49 years old) must have a pregnancy study within 7 days before starting treatment and the results are negative; Fertile patients must agree to use effective contraceptive measures to ensure that they are not pregnant during the study period and within 3 months after stopping treatment.

Exclusion Criteria:

1. Patients with central nervous system (CNS) metastasis or active CNS injury (i.e., imaging instability and symptomatic injury) (except patients with a single metastatic focus who are stable after treatment);
2. Within 4 weeks before the start of cell infusion, those who have received other anti-tumor treatments, taken corticosteroids (or analogues) or used systemic treatments that affect the immune system;
3. Blood pregnancy test positive or lactating female patients;
4. Uncontrolled accompanying diseases and active infectious diseases;
5. Patients who need anticoagulant therapy (warfarin or heparin);
6. The patient was allergic to naproxen, ibuprofen, trimetazidine/sulfamethoxazole and ampicillin.
7. Have a history of bone marrow transplantation or organ transplantation.
8. Patients who have previously used gene therapy drugs;
9. Patients with the following previous diseases or accompanying diseases:a) Patients who have been diagnosed as serious autoimmune diseases need systemic immunosuppressants (steroids) for a long time (more than 2 months) or immune-mediated symptomatic diseases, including ulcerative colitis, Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus (SLE) and autoimmune vasculitis (for example, Wegener's granulomatosis;b) Patients previously diagnosed with motor neuron disease caused by autoimmune disease; c) Patients with toxic epidermal necrolysis (TEN) in the past; d) Patients suffering from any mental illness, including dementia and mental state changes, which may affect informed consent and the understanding and performance of relevant questionnaires;e) It is determined that patients with serious uncontrollable diseases may be affected by this study; f) Patients with active malignant tumors such as basal or squamous skin cancer, superficial bladder cancer and breast cancer in situ in the past 5 years who have been completely cured and do not need follow-up treatment are not included;
10. Patients who have used immunotherapy for cancer in the past 6 months include: CIK, DC, DC-CIK, LAK and other lymphocyte-based immunotherapy patients;
11. Active/chronic human immunodeficiency virus (HIV), syphilis serological positive, active hepatitis B (hepatitis B surface antigen (HBsAg) positive and hepatitis B virus (HBV) deoxyribonucleic acid (DNA) > 500IU/ml or the lower detection limit of the research center [only when the lower detection limit of the research center is higher than 500 iu/ml]), or hepatitis C virus antibody positive;
12. Have a clear history of drug allergy or an allergic constitution; Patients participating in other clinical trials at the same time Other circumstances in which the researcher thinks that the patient should not participate in this experimental study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients (≥18 years old) HPV positive advanced cervical cancer (refer to FIGO standard)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
The objective remission rate assessed by the independent review committee according to RECIST1.1. | The time from the first administration to the first observation of disease recurrence or death of the patient was evaluated for up to 36 weeks.
  Main efficacy indicators

SECONDARY OUTCOMES:
Disease control rate (DCR) | The percentage of subjects who reached CR, PR and SD after treatment was analyzed.No more than 36 weeks.
  Secondary efficacy indicators
Progression-free survival (PFS) | The time interval between the patient's first treatment and the first record of disease progression or death.No more than 36 weeks.
  Secondary efficacy indicators

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, doctor, Study Director — Self
Locations (1):
- Wuxi People's Hospital, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No